CLINICAL TRIAL: NCT01265316
Title: Pediatric CPR Quality: Quantitative Measurement of Pediatric Cardiopulmonary Resuscitation (CPR) Quality During In-Hospital Cardiac Arrest
Brief Title: Measurement of the Quality of Pediatric CPR
Acronym: PediQ-CPR
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Highway Traffic Safety Administration (NHTSA) (U.S. Federal Agency); Laerdal Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: 10-007676
Record Dates: First submitted 2010-12-21; First posted 2010-12-23 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-02

CONDITIONS: Cardiac Arrest
Keywords: Cardiac arrest, CPR, pediatric
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: There is no intervention for this study. — There is no intervention for this study. The pre-NSR IDE for this study is simply a modification to allow for recording of data without intervention.

SUMMARY:
Outcomes for pediatric cardiopulmonary resuscitation (CPR) are suboptimal. CPR quality is directly related to resuscitation outcome, yet numerous deficiencies in CPR quality have been documented in adult studies. While similar deficiencies can be expected in pediatric resuscitation attempts, there is little to no data evaluating the existing quality of CPR performed during resuscitation attempts. Therefore, the objective of this study is to quantitatively evaluate existing CPR quality using a Q-CPR compression sensor manufactured by Philips Medical Systems with technology from Laerdal Medical.

DETAILED DESCRIPTION:
In the event of a cardiac arrest in the pediatric intensive care unit, a 24 hour paging system will notify the Cardiac Arrest Research Team to facilitate data collection. This system has been active as part of The Children's Hospital of Philadelphia (CHOP) Institutional Review Board (IRB) Protocol No. 2006-6-4839, and has resulted in capture of more than 95% of eligible events.

Cardiac arrest events requiring chest compressions in the PICU (pediatric intensive care unit) involving children greater than or equal to 1 year of age, but less than 8 years of age and who were previously screened, identified, and who have provided written consent are eligible for study. CPR quality will be recorded with the modified Heartstart MRx with Q-CPR Option, an external defibrillator with a chest compression sensor interposed between the hands of the rescuer providing chest compressions and the sternum of the patient. The device to be used is a regular Heartstart MRx with Quality of CPR (Q-CPR) Option cleared under 510(k) Premarket notification - K051134, but which has been modified for this study. In its current version, Q-CPR Option is approved for patients ≥ 8 years of age and has been utilized in the CHOP Pediatric Intensive Care Unit (PICU) under CHOP IRB Protocol No. 2006-6-4839. This Q-CPR Option on the Heartstart MRx has been modified for this study to accommodate children 1 year to less than 8 years of age. Since the device has been modified for use in this study, the device is an Investigational Device during this study regulated by the IDE regulation (CFR 21 Part 812). FDA has determined through a pre-investigational device exemption (IDE) process (I090674) that the use of the Heartstart MRx with the modified Q-CPR Option in a non-significant risk (NSR) device study. Two primary modifications were done on the Q-CPR Option: 1) changing the size of the compressions sensor footprint that interfaces with the patient's chest and 2) disabling the audiovisual Q-CPR feedback. Specifically the contact area of the compression sensor has been reduced to better mimic the area of the heel of a hand - the current recommended interface between the CPR administrator and the patient's chest during usual CPR / resuscitative care. Furthermore, no audiovisual feedback will be provided for this patient group as absolute measurement-based CPR quality targets do not exist for this age group. The device records CPR parameters (depth and rate of chest compressions), as well as electrocardiographic (ECG) data, and defibrillation shock data (if used). The pad relays this information to a recording component on the defibrillator which stores such data onto an internal data card. Once the cardiac arrest is completed, the MRx data can be exported to an external data card and downloaded to a secure laptop.

The investigator will use the Study Data Collection Form I in the Appendix to collect additional information immediately after resuscitation event has concluded. The patient's medical record will also be accessed and data will be collected as specified in the Medical Record Data Collection Form II. In addition to medical information, data collected will also include the post arrest chest depth in centimeters (cm) of the patient, chest circumference (cm) and details of the mattress and bed on which the child was resuscitated. Phase 2 procedures will be identical to those employed as per CHOP IRB Protocol No. 2006-6-4839.

ELIGIBILITY:
Inclusion Criteria:

Cardiac Arrest Inclusion Criteria

1. Cardiac arrests (chest compression events) occurring in the pediatric intensive care unit
2. Arrest patient age 1 year to less than 8 years
3. Subject pre-screened by a member of the Cardiac Arrest Research Team for safe use of the modified MRx/Quality of CPR (Q-CPR)
4. The modified MRx/Quality of CPR (Q-CPR) Compressions Sensor deployed

   Clinical Staff Inclusion Criteria
5. All clinical staff who participate in enrolled resuscitation events and who provided chest compressions

Exclusion Criteria:

Cardiac Arrest Exclusion Criteria

1. Cardiac arrests for patients classified as do not attempt resuscitation (DNAR)
2. Patient condition or size resulting in attending physician or physician fellow designee deciding not to deploy the modified MRx/Quality of CPR (Q-CPR) chest compression sensor (e.g., recent sternotomy)

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Cardiac arrests (chest compression events) occurring in the pediatric intensive care unit having consented for enrollment in the study.
Sampling Method: Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2010-10; Primary Completion 2013-01 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Determine the existing quality of CPR performed during the resuscitation of children 1year to less than 8 years of age. | 2 years

SECONDARY OUTCOMES:
Determine the chest wall stiffness of children in order to improve quantitative CPR modeling efforts and to facilitate the construction of more biofidelic pediatric manikins for CPR simulation and test dummies for automotive safety. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Vinay Nadkarni, MD, MS, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States